CLINICAL TRIAL: NCT00003648
Title: The Familial Colorectal Neoplasia Collaborative Group
Brief Title: Genetic Study of Patients and Families With a History of Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCCTG-974655; CDR0000066737 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-10-29 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Gene Rearrangement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and tumor samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients, family members, and control individuals complete an extended telephone interview, an extended personal interview, and an epidemiological survey, and contribute a blood specimen. Blood and tumor specimens are examined for the specific pattern of immunohistochemical expression of hMSH2 and HMLH1 to determine the frequency or lack of expression of these two protein products. Patients may be contacted periodically (about every 3 years) to update information about health, health practices, and family history. Patients do not receive the results of the genetic testing and the results do not influence the type or duration of treatment.
  Interventions: Genetic: DNA stability analysis; Genetic: gene rearrangement analysis

INTERVENTIONS:
Genetic: DNA stability analysis
Genetic: gene rearrangement analysis

SUMMARY:
RATIONALE: Determination of genetic markers for colorectal cancer may help doctors to identify patients who are at risk.

PURPOSE: Genetic testing study of patients and families with a history of colorectal cancer to identify patients who are at risk of developing colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Select patients with colon cancer and families at high-risk for colon cancer and collect leukocyte DNA, immortalized cell lines, plasma, and tumor specimens from these individuals and from control individuals. II. Develop patient education, counseling, and follow up plans for these individuals. III. Compare the frequency of defective DNA mismatch repair in individuals with familial colon cancer versus all colon cancers by using antibodies to the hMSH2 and hMLH1 protein products.

OUTLINE: This is a multicenter study. Patients, family members, and control individuals complete an extended telephone interview, an extended personal interview, and an epidemiological survey, and contribute a blood specimen. Blood and tumor specimens are examined for the specific pattern of immunohistochemical expression of hMSH2 and HMLH1 to determine the frequency or lack of expression of these two protein products. Patients may be contacted periodically (about every 3 years) to update information about health, health practices, and family history. Patients do not receive the results of the genetic testing and the results do not influence the type or duration of treatment.

PROJECTED ACCRUAL: At least 500-600 families (approximately 1500 patients) and the same number of matched controls will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Primary colorectal cancer and participating in one of the following NCCTG protocols: NCCTG-784852: No Treatment Control Versus Levamisole Versus Levamisole Plus 5-Fluorouracil NCCTG-794604: No Treatment Control Versus 5-FU by Portal Vein Infusion NCCTG-794751: Postoperative Radiation Versus Postoperative Radiation Plus Sequential Chemotherapy with Methyl CCNU and 5-FU NCCTG-844652: An Intergroup Study - An Evaluation of Levamisole Alone or Levamisole Plus 5-Fluorouracil as Surgical Adjuvant Treatment for Resectable Adenocarcinoma of the Colon NCCTG-864751: Phase III Protocol for Surgical Adjuvant Therapy of Rectal Carcinoma: A Controlled Evaluation of (A) Protracted-Infusion-5-Fluorouracil (5-FU) as a Radiation Enhancer and (B) 5-FU Plus Methyl-CCNU Chemotherapy NCCTG-874651: M/N - A Controlled Evaluation of Recombinant Interferon-Gamma (IFN-GM) and 5-FU and Folinic Acid With or Without Levamisole as Adjuvant Treatment for Resectable Adenocarcinoma of the Colon NCCTG-894651: A Controlled Phase III Evaluation of 5-Fluorouracil with Levamisole and Leucovorin as Adjuvant Treatment for Resectable Colon Cancer NCCTG-914653: A Phase III Evaluation of High-Dose Levamisole Plus 5-Fluorouracil and Leucovorin as Surgical Adjuvant Therapy for High-Risk Colon Cancer Adequate tissue for review OR Families of patients meeting the above criteria OR Colon cancer patient and population controls not in a high-risk family OR Spouse of a high-risk colon cancer patient

PATIENT CHARACTERISTICS: Age: Not specified Performance status: See Disease Characteristics Life expectancy: See Disease Characteristics Hematopoietic: See Disease Characteristics Hepatic: See Disease Characteristics Renal: See Disease Characteristics

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with colorectal cancer previously enrolled on NCCTG-784852, NCCTG-794751, NCCTG-844652, NCCTG-874651, NCCTG-894651, or NCCTG-914653.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 1998-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
frequency of defective DNA mismatch repair in individuals with familial colon cancer versus all colon cancers by using antibodies to the hMSH2 and hMLH1 protein products | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Noralane M. Lindor, MD, Study Chair — Mayo Clinic
Locations (12):
- United States (11):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada